CLINICAL TRIAL: NCT05127642
Title: Hemostatic Assessment of Postpartum Hemorrhage Cases Using Sonoclot Signature
Brief Title: Hemostatic Assessment of Postpartum Hemorrhage Using Sonoclot Signature
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rehab Abdelnasser Mohammed Omran, resident doctor, clinical Pathology department., Assiut University
Other Study IDs: HAOPPHCUSS
Record Dates: First submitted 2021-10-26; First posted 2021-11-19 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Postpartum hemorrhage patients
- Controls (non postpartum hemorrhage patients)

SUMMARY:
Postpartum hemorrhage is the leading cause of maternal morbidity and mortality throughout the world. Rapid diagnosis and early management improve maternal prognosis.

Postpartum hemorrhage is defined by a blood loss exceeding 500 ml during the 24 h after delivery.

There are many causes of postpartum hemorrhage. Most cases develop from uterine atony, which accounts for 75% of cases. Even though there are risk factors for postpartum hemorrhage, it is still an unpredictable obstetric emergency.

Coagulation plays an important role in postpartum hemostasis. Primary and especially secondary coagulation disorders are risk factors for Postpartum hemorrhage.

When bleeding occurs, the decrease in fibrinogen levels is the most rapid change observed among markers of coagulation. Recent studies show that fibrinogen concentration during the initial management of Postpartum hemorrhage is the most informative biological marker for the severity of the hemorrhage.

Various methods are used to record coagulation profile. One of them is estimation by sonoclot.

Viscoelastic hemostatic assays devices (such as sonoclot) have practical advantages as point-of-care devices for monitoring major hemorrhage including a set of parameters that assesses a global coagulation profile like fibrinogen and platelet count.

Identification of coagulopathy by viscoelastic point-of-care testing can be helpful in guiding management of Postpartum hemorrhage and preventing severe maternal outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. patients in childbearing period.
2. Patients with bleeding occurring in the first 24 hours after delivery (primary postpartum hemorrhage).
3. Patients with causes of Postpartum hemorrhage like uterine atony, preeclampsia, blood diseases as inherited and prepartum acquired coagulopathies, and others e.g., acute fatty liver of pregnancy, amniotic fluid embolism, etc.

Exclusion Criteria:

1. Patients with bleeding after 24 hours from delivery (secondary postpartum hemorrhage).
2. Patients with miscarriages (bleeding before 22 weeks of gestation) or Antepartum hemorrhage.
3. Traumatic causes of postpartum hemorrhage e.g., rupture uterus, abruptio placenta, Lacerations, hematomas, Uterine inversion, and iatrogenic trauma.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will be conducted in Assiut University Hospital, both clinical pathology department and obstetric and gynaecological department.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Haemostatic assessment in Postpartum haemorrhage Patients using Sonoclot signature. | 3 years

REFERENCES:
- [Result] Liew-Spilger AE, Sorg NR, Brenner TJ, Langford JH, Berquist M, Mark NM, Moore SH, Mark J, Baumgartner S, Abernathy MP. Viscoelastic Hemostatic Assays for Postpartum Hemorrhage. J Clin Med. 2021 Aug 31;10(17):3946. doi: 10.3390/jcm10173946. PMID 34501395
- [Result] Huissoud C, Carrabin N, Audibert F, Levrat A, Massignon D, Berland M, Rudigoz RC. Bedside assessment of fibrinogen level in postpartum haemorrhage by thrombelastometry. BJOG. 2009 Jul;116(8):1097-102. doi: 10.1111/j.1471-0528.2009.02187.x. Epub 2009 May 12. PMID 19459866
- [Result] Gallos ID, Williams HM, Price MJ, Merriel A, Gee H, Lissauer D, Moorthy V, Tobias A, Deeks JJ, Widmer M, Tuncalp O, Gulmezoglu AM, Hofmeyr GJ, Coomarasamy A. Uterotonic agents for preventing postpartum haemorrhage: a network meta-analysis. Cochrane Database Syst Rev. 2018 Apr 25;4(4):CD011689. doi: 10.1002/14651858.CD011689.pub2. PMID 29693726
- [Result] Henriquez DDCA, Bloemenkamp KWM, van der Bom JG. Management of postpartum hemorrhage: how to improve maternal outcomes? J Thromb Haemost. 2018 Jun 8. doi: 10.1111/jth.14200. Online ahead of print. PMID 29883040
- [Result] Cortet M, Deneux-Tharaux C, Dupont C, Colin C, Rudigoz RC, Bouvier-Colle MH, Huissoud C. Association between fibrinogen level and severity of postpartum haemorrhage: secondary analysis of a prospective trial. Br J Anaesth. 2012 Jun;108(6):984-9. doi: 10.1093/bja/aes096. Epub 2012 Apr 6. PMID 22490316
- [Result] Benes J, Zatloukal J, Kletecka J. Viscoelastic Methods of Blood Clotting Assessment - A Multidisciplinary Review. Front Med (Lausanne). 2015 Sep 14;2:62. doi: 10.3389/fmed.2015.00062. eCollection 2015. PMID 26442265
- [Result] Curry NS, Davenport R, Pavord S, Mallett SV, Kitchen D, Klein AA, Maybury H, Collins PW, Laffan M. The use of viscoelastic haemostatic assays in the management of major bleeding: A British Society for Haematology Guideline. Br J Haematol. 2018 Sep;182(6):789-806. doi: 10.1111/bjh.15524. Epub 2018 Aug 2. No abstract available. PMID 30073664